CLINICAL TRIAL: NCT01609179
Title: IPI-926 Extension Protocol for Continuation of IPI-926 Treatment in Patients Experiencing Clinical Benefit While Enrolled in an IPI-926 Protocol
Brief Title: IPI-926 Extension Protocol for Continuation of Treatment With IPI-926
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Infinity Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPI-926-09
Record Dates: First submitted 2012-05-29; First posted 2012-05-31 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Basal Cell Carcinoma; Chondrosarcoma
MeSH Terms: conditions — Carcinoma, Basal Cell; Chondrosarcoma | interventions — IPI-926

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IPI-926 (Experimental)
  Interventions: Drug: IPI-926

INTERVENTIONS:
Drug: IPI-926 — IPI-926 is administered orally as a capsule formulation, as a fixed dose in mg/day. Patients will be administered the same dose with same cycle length of IPI-926 and combination therapy that they were receiving in the original protocol at the time of transition into the extension study. The following are potential once-daily doses that patients are receiving in original protocols: 60 mg, 90 mg, 100 mg, 110 mg, 130 mg, or 160 mg.
  Other Names: saridegib

SUMMARY:
A treatment protocol that enables patients to have continued access to IPI-926.

DETAILED DESCRIPTION:
The extension protocol is a continuation of treatment with IPI-926, as administered to each individual patient during participation in their original IPI-926 protocol.

Patients who are completing their participation in the original IPI-926 protocol in which they enrolled, as defined in the original protocol, and, have stable disease or confirmed complete or partial response as defined by the original protocol may continue to receive treatment with IPI-926 in the extension protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form
2. Currently receiving IPI-926 while participating in an Infinity-sponsored IPI-926 study. Note: For blinded studies, patient's treatment assignment must be unblinded according to the instructions in the original protocol to confirm they are receiving IPI-926.
3. Eastern Cooperative Oncology Group (ECOG) performance status: 0 or 1.
4. Documented response or stable disease, as defined in the original protocol, at the time of entry to the extension study.
5. Willingness and ability to continue IPI-926 dispensation and follow-up procedures at the current investigational site.
6. Willingness and ability to comply with scheduled visits, treatment plans, and laboratory tests and other study procedures.
7. Women of child-bearing potential (WCBP), defined as a sexually mature woman who has not undergone a hysterectomy or tubal ligation or who has not been naturally postmenopausal for at least 24 consecutive months, must have a negative serum or urine pregnancy test prior to treatment. All WCBP, all sexually active male patients, and all partners of patients must agree to use adequate methods of birth control throughout the study.

Exclusion Criteria:

1. Discontinued IPI-926 or withdrew informed consent to participate in original Infinity-sponsored IPI-926 study.
2. Require addition of or change to a new concomitant therapy to adequately treat the malignancy under study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-03; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs), and laboratory test results | Up to 30 days after the last patient study visit
  Monitoring of AEs, including SAEs as well as review of laboratory sample test data to assess safety and tolerability of IPI-926

CONTACTS AND LOCATIONS:
Overall Officials: Tess Schmalbach, MD, Study Director — Infinity Pharmaceuticals, Inc.
Locations (2):
- United States (2):
  - University of Colorado Denver, Aurora, Colorado
  - Johns Hopkins, Baltimore, Maryland